CLINICAL TRIAL: NCT02372864
Title: PURSUE - Psychosexual Consequences of Risk-reducing Salpingooophorectomy in BRCA1/2 Mutation Carriers
Brief Title: Psychosexual Consequences of Risk-reducing Salpingo-oophorectomy
Acronym: PURSUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Catheleine van Driel, MD/PhD candidate, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PURSUE2014
Record Dates: First submitted 2015-02-11; First posted 2015-02-26 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Cancer
Keywords: Ovariectomy; Mindfulness; Postmenopause; Hot Flashes
MeSH Terms: conditions — Ovarian Neoplasms; Hot Flashes | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care as usual (No Intervention): All participants in the intervention and control group receive the care as usual. The care as usual consists of a clinic appointment with the research nurse. In this appointment the RRSO-induced menopausal complaints will be discussed in more detail. Depending on the complaints at hand, information, reassurance and life style advice will be offered. A leaflet with relevant information will be provided for. Furthermore, the usual medical care may include prescription of (non-)hormonal medicationsTwelve weeks after the clinic appointment, the research nurse will contact all participants per telephone to ask whether there are issues that remain to be addressed.
  Participants are allowed to continue the use of all their current medication.
- Mindfullness based stress reduction (Experimental)
  Interventions: Behavioral: Mindfulness based stress reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction (MBSR) — Mindfulness based stress reduction (MBSR) is a standardized eight-week psychosocial intervention delivered by certified trainers. The programme consists of a weekly class of two and half hours for a period of eight weeks and a full retreat day. Furthermore participants are asked to practice exercises at home for 45 minutes, six days a week. The MBSR class will consist of ten to twelve persons, starting at different weekdays and moments of the day. If during the inclusion process it becomes apparent that a group of participants (provided a sufficient group size) comes from a region (e.g. Friesland or Overijssel) with a considerable amount of traveling time to the UMCG, efforts will be made to start a MBSR training in the region with trainers from the UMCG.
  Arms: Mindfullness based stress reduction

SUMMARY:
Short Rationale: Risk-reducing salpingo-oophorectomy (RRSO) is a mainstay in preventing ovarian cancer in BRCA1/2 mutation carriers, as ovarian cancer screening is ineffective in detecting ovarian cancer in an early and curable stage. Women who underwent RRSO experienced bothersome menopausal symptoms and worsening of sexual functioning related to acute surgical menopause. Hormone replacement therapy (HRT) will mitigate some of the RRSO induced menopausal complaints, however it does not reduce the complaints to a premenopausal level and the sexual symptoms are not alleviated. Mindfulness interventions were found to improve sexual functioning and alleviate menopausal symptoms in various populations. It has not been investigated whether mindfulness-based stress reduction (MBSR) is effective in mitigating the RRSO-induced menopausal complaints in BRCA1/2 mutation carriers and if this effect is sustained over a longer period of time.

Objective: To examine the effect of MBSR training on the menopause-specific quality of life in BRCA1/2 mutation carriers who experience RRSO-induced menopausal complaints.

Study population: Female BRCA1/2 mutation carriers who were younger than 52 years at the time of RRSO reporting two or more moderate to severe menopause related complaints after undergoing RRSO.

Study design: Prospective randomized controlled trial with a follow-up time of twelve months conducted at the University Medical Center Groningen (UMCG)

Intervention: Eight-week MBSR training consisting of a weekly class of two and half hours and a full retreat day. Furthermore participants are asked to practice mindfulness exercises at home for 45 minutes, six days a week.

Main study parameters/endpoints: Menopause specific quality of life score measured by the Menopause-specific quality of life questionnaire (MENQOL). Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no risks associated with taking part in a MBSR training or filling out the questionnaires that will be used in this study. The content of the questionnaires concerns intimate matters and could be considered burdensome. A possible benefit for the participants of the MBSR training is that participants will be more able to cope with their complaints after RRSO. The group relatedness is reflected in the fact that RRSO is specifically performed in women with a hereditary risk of ovarian cancer such as BRCA1/2 mutation carriers.

DETAILED DESCRIPTION:
OBJECTIVES This study will evaluate the effectiveness of a mindfulness-based intervention in alleviating RRSO-induced menopausal complaints in BRCA1/2 mutation carriers. The intervention to be tested is MBSR training. The investigators hypothesize that women in the MBSR group will report statistically significantly greater improvement of menopause-specific quality of life from baseline to twelve weeks when compared to the control group and that this improvement will be maintained at six months and twelve months. The investigators also hypothesize that women in the MBSR group will report a statistically significantly greater improvement in sexual functioning and a decrease in sexual distress from baseline to twelve weeks when compared to the control group and that this improvement will be maintained at six and twelve months.

The primary objective is to examine the effect of MBSR training on the menopause-specific quality of life in BRCA1/2 mutation carriers who experience RRSO-induced menopausal complaints.

The secondary objective is to examine the effect of MBSR training on sexual functioning and distress in BRCA1/2 mutation carriers who experience RRSO-induced menopausal complaints.

STUDY DESIGN The study is a prospective, randomized controlled trial, with an intervention group that receives an eight-week MBSR training as well as care as usual and a control group that only receives care as usual. All participants will be asked to fill out questionnaires regarding menopausal and sexual complaints at baseline before randomization (T0) and at twelve weeks (T1), six (T2) and twelve months (T3) after randomization. The study will be conducted at the family cancer clinic of the UMCG.

STATISTICAL ANALYSIS The two treatment arms will be summarized at baseline with frequencies for categorical variables and means, ranges and SDs for continuous variables. Scores for the MenQOL, FSFI and FSDS will be calculated according to published scoring algorithms.

A linear mixed effects analysis will be performed on the relationship between the MenQOL score and the intervention. The scores on the MenQOL at 12 weeks, 6 months and 12 months will be modelled as a function of treatment arm, time moment, their interaction. An unstructured correlation matrix will be assumed, unless the data indicate the presence of another correlation structure. If the groups are unbalanced, covariates will added to the model. All analysis will be conducted on an intention-to-treat basis. All analyses will be performed with SPSS.

Similar analyses will be conducted for the FSFI and FSDS, which will be used as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* younger than 52 years at the time of risk-reducing salpinghoophorectomy
* no active cancer

Exclusion Criteria:

* severe cognitive or psychiatric problems
* no sufficient mastery of the Dutch language

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the menopause-specific quality of life questionnaire (MENQOL) score. | Baseline, 12 weeks, 6 and 12 months
  The MENQOL is a self-administered 29-item questionnaire developed to assess quality of life in menopausal women. It not only records menopausal symptoms, but also the degree of bother women experience due to the menopausal symptoms. It consists of four domains: vasomotor (three items), psychosocial (seven items), physical (sixteen items) and sexual (three items). All items firstly ask whether or not a woman has experienced the item in the prior four weeks. If this was the case she is then asked to indicate how much she was bothered on a zero (no bother) to seven (extreme bother) scale. Higher scores on the MENQOL reflect a poorer menopause-specific quality of life. The minimal clinically important difference was found to be 1.0. The MENQOL is available in Dutch and has undergone extensive linguistic validation.

SECONDARY OUTCOMES:
Change from baseline in the female sexual function index questionnaire (FSFI) score. | Baseline, 12 weeks, 6 and 12 months
  FSFI is a self-report questionnaire widely used to assess sexual functioning. It consists of nineteen items and the following six sub-domains: desire (items 1 and 2), arousal (items 3-6), lubrication (items 7-10), orgasm (items 11-13), satisfaction (items 14-16) and pain (items 17-19). Each domain can be scored from zero to five on a Likert-type scale. The higher the scores are the better the sexual functioning has been in the prior four weeks. As a clinical cutoff score for sexual dysfunction 26.55 is used. The FSFI is available in Dutch and has undergone extensive linguistic validation
Change from baseline in the female sexual distress scale (FSDS) score. | Baseline, 12 weeks, 6 and 12 months
  The FSDS is a self-report questionnaire that is used to assess sexual activity related distress in four weeks prior to adminstration. The FSDS consists of twelve items and can be scored on a five point Likert-type scale from zero to four and has a maximum total score of 48. A score of fifteen or higher is the cutoff score for clinically significant distress. The FSDS is available in Dutch and has undergone extensive linguistic validation

CONTACTS AND LOCATIONS:
Overall Officials: Marian JE Mourits, prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands